CLINICAL TRIAL: NCT05791136
Title: Toripalimab After Radiotherapy Alone in Elderly Esophageal Squamous Cell Carcinoma: A Prospective Phase II Clinical Trial
Brief Title: Immunotherapy After Radiotherapy in Elderly ESCC
Acronym: TREE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Central Hospital of Lishui City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJLSRT-001
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Esophageal Squamous Cell Carcinoma by AJCC V8 Stage
Keywords: Esophageal Squamous Cell Carcinoma; PD-1; Elderly; Radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; toripalimab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Sequential Toripalimab (Experimental): Radiotherapy:Intensity-modulated radiotherapy (IMRT) Immunotherapy: Toripalimab
  Interventions: Radiation: Radiotherapy; Drug: Toripalimab

INTERVENTIONS:
Radiation: Radiotherapy — 95% PGTV56-60Gy/28-30 fractions, 2Gy/1 fractions; 95% PTV50.4-54Gy/28-30 fractions, 1.8Gy/1 fractions; 5 days a week; 6 weeks.
  Other Names: Intensity-modulated radiotherapy (IMRT)
Drug: Toripalimab — Toripalimab (200 mg, intravenously infused) will be administered as the maintenance treatment every 3 weeks within 4 weeks after the completion of radiotherapy for 1 years or until progression, intolerable toxicity, or physician/patient decision
  Other Names: Immunotherapy

SUMMARY:
The incidence and mortality of esophageal squamous cell carcinoma are at the forefront in China.Most part of patients are elderly. Concurrent chemoradiotherapy is the standard treatment for unresectable locally advanced esophageal squamous cell carcinoma. Most elderly patients cannot tolerate concurrent chemotherapy because of complications and other reasons. Immunotherapy has definite efficacy and low toxicity in advanced esophageal squamous cell carcinoma, and the results combined with radiotherapy have also been preliminarily reported. Therefore, it is necessary to further explore the efficacy and safety of radiotherapy combined with immunotherapy in elderly patients with esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm, phase Ⅱ clinical study to evaluate the efficacy and safety of radiotherapy alone followed by sequential injection of Toripalimab in elderly patients with unresectable esophageal squamous cell carcinoma who could not accept concurrent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥75 years old, regardless of gender；
2. Esophageal cancer confirmed by histology or cytology；
3. Unresectable, unable to tolerate or refuse surgery and concurrent chemoradiotherapy；
4. Unable to tolerate chemotherapy；
5. There are at least one lesions measurable according to RECIST 1.1；
6. Stage II-iva (AJCC 8 TNM classification)
7. Endoscopic ultrasonography confirmed that esophageal lesions did not invade adjacent organs (T1-4a).；
8. ECOG PS 0-1；
9. Forced expiratory volume (FEV) >0.8 liter；
10. Life expectancy of at least 12 weeks；
11. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, biotherapy，etc.
12. Has sufficient organ function： (1) Blood routine: ANC≥1.5×109/L; PLT≥50×109/L; HGB≥90 g/L((No blood transfusion and blood products within 14 days, no use of G-CSF and other blood-stimulating factors to correct)) (2) Liver function: TBIL ≤ 1.5 × ULN，ALT、AST ≤2.5 × ULN， (3) Renal function: Cr≤1×ULN or crcl ≥50 ml/min (4) Adequate haemostasis laboratory data prior to randomization: INR or PT ≤1.5×ULN (If the subject was receiving anticoagulant therapy, as long as the PT was within the intended use range of anticoagulant drugs) (5) Myocardial enzymes were within the normal range.
13. Patients voluntarily joined this study, signed informed consent and provided diagnosis and treatment data after cancer diagnosis before entering the group, good compliance, and cooperation with follow-up visits;

Exclusion Criteria:

1. Synchronous or metachronous second primary malignancy. Participants with basal cell carcinoma of the skin, or cervical cancer in situ that have undergone potentially curative therapy are not excluded from the study;
2. with multifocal primary esophageal cancer;
3. The pathological diagnosis was esophageal small cell carcinoma, adenocarcinoma, or mixed carcinoma.
4. Esophageal squamous cell carcinoma with active bleeding within 2 months of the primary lesion；
5. Patients whose imaging has shown that the tumor has invaded the important blood vessels or the investigator judges that the tumor is likely to invade the important blood vessels and cause fatal hemorrhage during the follow-up study
6. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, glomerulonephritis, thyroiditis (patients with vitiligo or asthma has been completely relieved in childhood, and do not need any intervention during adulthood can be included; patients with type I diabetes with good insulin control can also be included; hypothyroidism caused by autoimmune thyroiditis requiring hormone replacement therapy can also be included)
7. Clinically significant cardiac disease or impaired cardiac function, such as: MeanQT interval corrected for heart rate (QTc) ≥470 ms, Congestive heart failure requiring treatment (New York Heart Association [NYHA] grade > 2), left ventricular ejection fraction (LVEF) <50% as determined by Echocardiography.
8. Active infection or fever of unknown origin > 38.5 ° C during screening or before the first dose (tumor-related fever, as judged by the investigator, was eligible);
9. Current pneumonitis or interstitial lung disease or history of pneumonitis or interstitial lung disease.
10. Has had congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-DNA ≥ 104 copies/ml) or hepatitis C (HCR-RNA was higher than the detection limit of the analytical method);
11. Previous treatment with another PD-1, PD-L1；
12. Known hypersensitivity to macromolecular protein preparations or to any anti-PD-1 antibody component;；
13. Immunosuppressive drugs used within 7 days prior to the initial study treatment, excluding local glucocorticoids, or systemic glucocorticoids at physiological doses (i.e., no more than 10 mg/ day of prednisone or equivalent doses of other glucocorticoids); Systemic steroid doses of less than 10 mg of prednisone daily or its equivalent are allowed in patients receiving physiologic replacement steroid doses without autoimmune disease.
14. if they had undergone major surgery patients must have fully recovered from surgery with no major ongoing safety issues before the experiment begins.
15. Currently participating in an interventional clinical research treatment, or has received another investigational drug or used an investigational device within 4 weeks prior to the first administration of the drug.
16. Live vaccine within 4 weeks prior to first dose (Cycle 1, Day 1); NOTE: Injectable inactivated viral vaccine against seasonal influenza is allowed; however, live attenuated influenza vaccine for intranasal administration is not allowed.
17. The investigator considers it unsuitable for inclusion. Patients with uncontrollable seizures or loss of self-control due to mental illness. serious abnormal laboratory test results, family, or social factors, which may affect the safety of the subjects or the data collection.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  We aim to evaluate the progression-free survival (PFS) of elderly patients with unresectable esophageal squamous cell carcinoma who were unable to accept concurrent chemotherapy and received sequential treatment with Triptolide injection after radiotherapy alone.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  Overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence .
Objective response rate (ORR) | 2 years
  Objective response rate (ORR) is defined as the proportion of patients with a complete response(CR) or partial response(PR) to treatment according to RECIST v1.1.
Duration of response (DOR) | 2 years
  Duration of response (DOR) was determined from date of initial response to PD according to RECIST v1.1.
Time to death or distant metastasis (TTDM) | 2 years
  Time to death or distant metastasis (TTDM) according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Zhifeng Tian, M.D, Principal Investigator — Lishui Municipal Central Hospital，Zhejiang，China

IPD SHARING:
Plan to Share IPD: No
participant number,age,gender